CLINICAL TRIAL: NCT03347682
Title: Reliability and Construct Validity of the Turkish Version of the Prosthesis Donning and Doffing Questionnaire in Transtibial Amputees.
Brief Title: Turkish Validation of Prosthesis Donning and Doffing Questionnaire
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2017.659
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2017-10

CONDITIONS: Amputation; Traumatic, Leg, Lower
Keywords: Amputation, prosthesis,psychometrics, questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group: Transtibial amputees: After translation/retranslation of the Prosthesis donning and doffing questionnaire, transtibial amputees will be asked to complete a quality of life evaluation Nottingham Health Profile-NHP, a satisfaction evaluation Satisfaction with Prosthesis -SATPRO and the Turkish version of the Prosthesis donning and doffing questionnaire twice (1-3 days apart).
  Interventions: Other: Satisfaction with Prosthesis -SATPRO; Other: Nottingham Health Profile-NHP; Other: Prosthesis donning and doffing questionnaire

INTERVENTIONS:
Other: Satisfaction with Prosthesis -SATPRO — questionnaire 1
Other: Nottingham Health Profile-NHP — questionnaire 2
Other: Prosthesis donning and doffing questionnaire — questionnaire 3

SUMMARY:
The aim of this study is to investigate the Reliability and construct validity of the Turkish version of the Prosthesis donning and doffing questionnaire in transtibial amputees.

DETAILED DESCRIPTION:
Knowing that a socket and suspension system should be donned and doffed few times during the day and night, it is important to measure ease of donning and doffing. Effortless donning and doffing does appear to have a posi- tive effect on satisfaction with a prosthesis. The socket and suspension systems require different methods of don and doff, some of which are time-consuming and necessi- tate more hand strength and cognitive effort than others. The pin/lock suspension needs few re-adjustments of residual limb within the socket so that the pin is fully locked distally. The seal-in system, for example, needs a longer period as first the amputee needs to spray either the inner socket or the seals, and then remove the socket valve and push the limb into the socket and put back the valve. Instruments are available to evaluate socket comfort such as the socket comfort score, yet to the authors' knowledge no instrument has been developed that focuses on donning and doffing quality of prosthesis. The clearer the insight into suspension systems, the easier will be the selection for prosthetist.

There are different questionnaires in the fields of prosthetics and orthotics such as Prosthetic Evaluation Questionnaire (PEQ), Trinity Amputation and Prosthesis Experience Scales (TAPES), Orthotic Prosthetic User's Survey (OPUS), Houghton scale of prosthetic use, and Amputee Body Image Scale (ABIS) However, few of these instruments address donning and doffing of prosthesis. There is no questionnaire in Turkish available to evaluate the donning and doffing procedures of suspension systems. Thus, the aim of this study is to investigate the Reliability and construct validity of the Turkish version of the Prosthesis donning and doffing questionnaire in transtibial amputees.

After obtaining permission from the developers of the Prosthesis donning and doffing questionnaire, the Turkish version of the instrument will be developed. For the translation process, established guidelines for patient reported outcome (PRO) instrument translation and include both forward and backward (reverse) translation of instructions, items, and response options by independent translators; review by bilingual experts; reconciliation of translations; and cognitive testing of the translated instruments, as described by Eremenco et al., 2005 or Reeve et al., 2013 were followed.The necessity of performing a cultural adaptation for the use of the Turkish version among Turkish amputees will be assessed. Level of education part of the manuscript is planned to be changed bacause it doesn't fit the education system in Turkey). After discussions between the study investigators and translators, a Turkish version of the Prosthesis donning and doffing questionnaire that corresponded as closely as possible to the original survey will be produced. Each subject will be asked to complete the Turkish version of the Prosthesis donning and doffing questionnaire twice (1-3 days apart). To evaluate the validity of the Turkish version of the Prosthesis donning and doffing questionnaire, the Nottingham Health Profile(NHP), Satisfaction with Prosthesis -SATPRO surveys will be used.

Satisfaction with the prosthesis has the following subscales: aesthetic satisfaction with the prosthesis, weight satisfaction with the prosthesis and functional satisfaction with the prosthesis. The weight satisfaction subscale has just one item, which is answered with a 5-point Likert-type scale, whereas both aesthetic satisfaction and functional satisfaction with prosthesis have five items, each answeredwith a 5-point Likert-type scale.

The Turkish version of Nottingham Health Profile(NHP), a generic quality of life measurement tool, has been showed to be a valid and reliable outcome measurement. For this reason it will be used to analyse the construct validity of the Prosthesis donning and doffing questionnaire. NHP (translated by Küçükdeveci et a.) includes the following six subdomains: energy level, physical activities, pain, sleep, emotional reaction and social isolation. The sum of the scores of each subdomain equals.12 The SATPro is a 15-item questionnaire that measures general satisfaction with a prosthesis. The Turkish version of the questionnaire, developed by Simsek, was used. Each item on the questionnaire is scored between 0 and 3.

ELIGIBILITY:
Inclusion Criteria:

Transtibial amputee, who used prosthesis for at least 1 year and had no cognitive disorders.

Exclusion Criteria:

1. Bilateral amputation or upper extremity amputation
2. Amputation levels other than transtibial
3. Cognitif impairement
4. Presence of neuroma, bony growths, skin lesions, wounds leading unability to use prosthesis.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Transtibial amputees aged 18-65 years and using their well fitted prosthesis at least 1 year
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Prosthesis donning and doffing questionnaire | Day 0
  Satisfaction was measured through Prosthesis donning and doffing questionnaire. The total score may be categorized into "low, moderate, and high" as follows-total score ⩽ 2: low; total score = 3 and 4: moderate; and total score ⩾ 5: high. The higher score may be interpreted as higher quality and satisfaction with the donning and doffing.
Prosthesis donning and doffing questionnaire | Day 3
  Satisfaction was measured through Prosthesis donning and doffing questionnaire. The total score may be categorized into "low, moderate, and high" as follows-total score ⩽ 2: low; total score = 3 and 4: moderate; and total score ⩾ 5: high. The higher score may be interpreted as higher quality and satisfaction with the donning and doffing.

SECONDARY OUTCOMES:
Satisfaction with Prosthesis -SATPRO | Day 0
  The questionnaire includes 15 items developed on the basis of the most significant criteria used by the person when selecting a technical aid. Minimum score 0 maximum score 45.
Satisfaction with Prosthesis -SATPRO | Day 3
  The questionnaire includes 15 items developed on the basis of the most significant criteria used by the person when selecting a technical aid. Minimum score 0-maximum score 45.
Nottingham Health Profile | Day 0
  The Nottingham Health Profile is intended for primary health care, to provide a brief indication of a patient's perceived emotional, social and physical health problems. The number of questions answered "yes" in each subgroup is divided by the total number of questions in the same subgroup and the result is multiplied by 100. Each subgroup has a value of between 0 and 100, with 100 points being considered the best general QoL for the calculated subgroup and 0 points being considered as the worst QoL for the same subgroup.
Nottingham Health Profile | Day 3
  The Nottingham Health Profile is intended for primary health care, to provide a brief indication of a patient's perceived emotional, social and physical health problems. The number of questions answered "yes" in each subgroup is divided by the total number of questions in the same subgroup and the result is multiplied by 100. Each subgroup has a value of between 0 and 100, with 100 points being considered the best general QoL for the calculated subgroup and 0 points being considered as the worst QoL for the same subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Giray Esra, MD, Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang M, Turner-Smith AR, Tanner A, Roberts VC. Clinical investigation of the pressure and shear stress on the trans-tibial stump with a prosthesis. Med Eng Phys. 1998 Apr;20(3):188-98. doi: 10.1016/s1350-4533(98)00013-7. PMID 9690489
- [Result] Abu Osman NA, Eshraghi A, Gholizadeh H, Wan Abas WAB, Lechler K. Prosthesis donning and doffing questionnaire: Development and validation. Prosthet Orthot Int. 2017 Dec;41(6):571-578. doi: 10.1177/0309364617690397. Epub 2017 Feb 13. PMID 28190376
- [Result] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Result] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Result] Kuru P, Akyuz G, Yagci I, Giray E. Hypovitaminosis D in widespread pain: its effect on pain perception, quality of life and nerve conduction studies. Rheumatol Int. 2015 Feb;35(2):315-22. doi: 10.1007/s00296-014-3099-7. Epub 2014 Aug 2. PMID 25085713
- [Result] Schaffalitzky E, Gallagher P, Maclachlan M, Wegener ST. Developing consensus on important factors associated with lower limb prosthetic prescription and use. Disabil Rehabil. 2012;34(24):2085-94. doi: 10.3109/09638288.2012.671885. Epub 2012 Apr 12. PMID 22494367
- [Result] Eshraghi A, Osman NA, Gholizadeh H, Karimi M, Ali S. Pistoning assessment in lower limb prosthetic sockets. Prosthet Orthot Int. 2012 Mar;36(1):15-24. doi: 10.1177/0309364611431625. Epub 2012 Jan 22. PMID 22269941